CLINICAL TRIAL: NCT00360139
Title: A Phase IV, Prospective, Non-Blinded, Non-Randomized, Single-Center Clinical Trial to Determine the Longevity, Duration, and Volume-Correcting Efficacy of Sculptra™ Dermal Filler for the Correction of Contour Deformities Caused by Lipoatrophy
Brief Title: Clinical Trial to Determine the Efficacy of Sculptra™ Dermal Filler for the Correction of Contour Deformities Caused by Lipoatrophy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc. (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLA-SCULP-0305
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Lipodystrophy; Emaciation
Keywords: Sculptra; lipoatrophy; emaciation; facial; dermal filler; poly-L-lactic acid; Dermik; SpaMD; Sanofi; Facial lipoatrophy; Facial emaciation
MeSH Terms: conditions — Lipodystrophy; Emaciation; Facies

INTERVENTIONS:
Device: Sculptra Injection

SUMMARY:
Lipoatrophy is a condition that affects certain individuals, most commonly those who are infected with the HIV virus. Lipoatrophy however can also affect individuals who suffer from recurrent systemic infections, those who have a weakened immune system, or certain patients who suffer from cancer or receive chemotherapeutics. In contrast, lipoatrophy can sometimes be present in individuals who are perfectly healthy but have genetically predisposing factors that can contribute to facial emaciation or lipoatrophy.

The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume. These often elastic contour fillers (also known as soft tissue augmentation devices) can correct hollowness around the eyes, add fullness to thin lips, balance a disproportionate face or correct topographical anomalies.

This study aims to:

* Objectively measure the improvement of contour-deformities after Sculptra™ injection from baseline to study closure by utilizing the Primos™ photographic/topographical measuring system.
* Evaluate the efficacy, longevity and duration of volume-correction in subjects which are both HIV positive and HIV negative.
* Assess the safety of Scupltra™ dermal filler when used to correct volume deformities caused by lipoatrophy in subjects that are HIV negative.

DETAILED DESCRIPTION:
Soft tissue fillers are used to temporarily fill facial lines and wrinkles and augment contour deformities. There are a variety of soft tissue fillers available.

Sculptra™ has been used to correct dermal atrophy in both the HIV and non-HIV populations. Almost all clinical trials have used a visual assessment scale to grade correction as well as persistence. Recently, dermal ultrasound has been used to provide an objective measurement of dermal thickening, but the ultrasound procedure measures only a fraction of the dermis and is subject to a high degree of variability because of the difficulty in measuring the same area. Our protocol utilizes the Primos ½ face system to produce a 3-dimensional evaluation of a large area. This will produce excellent reproducible results as well as outstanding photographs for patient demonstration.

Sculptra™ is an injectable implant that contains microparticles or poly-L-lactic acid, a biocompatible, biodegradable, synthetic polymer from the alpha-hydroxy-acid family. Sculptra™ is reconstituted prior to use by the addition of sterile water for injection, USP (SWFI) to form a sterile non-pyrogenic suspension.

Comparison:

Dermik's Vega Study - The Vega study was a 96-week, open-label, uncontrolled, single-center study to determine the treatment effects of Sculptra on the signs of lipoatrophy of the face in 50 patients infected with human immunodeficiency virus. Patients had a mean age of 45 years (range 33-58), 84% were Caucasian and 98% were male. All patients had little or no adipose tissue in cheek area at baseline, indicating severe facial lipoatrophy (mean adipose thickness of 0.5±0.7 mm, ranging from 0.0 to 2.1 mm).

Treatment injection sessions were conducted at approximately two-week intervals, and the majority (86%) of the patients received four to five injection sessions. Generally, one vial of product was injected intradermally into multiple points of each cheek at each injection session. The quantity of injected product and number of injection sessions depended upon the severity of the facial depression.

All patients experienced increases in skin thickness in the treatment area (minimum increase of 2.2 mm noted at Week 8 visit). Statistically significant increases above baseline values of mean skin thickness were noted at all time points (Weeks 8, 24, 48, 72 and 96) during the study. Increases in mean skin thickness changes above baseline persisted for up to 2 years.

This study follows the same general design as the Vega study.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral lipoatrophy corresponding to a visual grade 2 or above in the attached lipoatrophy scale.
2. Available and willing to attend all follow-up visits.
3. Age > 18 years.
4. Able and willing to give informed consent.

Exclusion Criteria:

1. Known allergy or sensitivity to Sculptra™, suture material or any material that in the investigator's opinion may cause an allergic reaction.
2. The subject has received a soft tissue augmentation to the area to be treated within the last 6 months.
3. Subject is unwilling to forgo any cosmetic augmentation procedures for the duration of the study.
4. The subject has received autologous fat transfer in the last 6 months.
5. Subject is suffering from facial Kaposi's sarcoma.
6. The subject has active skin diseases or inflammation on or near the area of injection, such as psoriasis, herpes zoster, infection, or discoid lupus.
7. History of sensitivity to lidocaine.
8. Pregnant or nursing. (Premenopausal or nonsurgically sterile women must have a negative urine pregnancy test and must be using an adequate method of birth control.)
9. Subject has ever received an injection or implant of silicone in the area to be treated.
10. Subject is currently on any metabolic augmentation medications such as anabolic steroids.
11. Current use of anticoagulant therapy or has a history of hemorrhagic disorders.
12. History of connective tissue disease or other related disorder that in the investigator's opinion excludes the subject from the study.
13. Subject is involved in any other research study involving an investigational product, or has concluded a study less than 30 days ago.
14. The subject is suffering from any medical condition or complication that in the investigator's opinion places the subject at risk by participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Study Completion 2008-12

PRIMARY OUTCOMES:
Volume correction and longevity of correction | at 12 and 24 months

SECONDARY OUTCOMES:
Safety in non-HIV positive subjects

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P. Goldman, M.D., Principal Investigator — Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc.
Locations (1):
- Dermatology Cosmetic Laser Associates of La Jolla, La Jolla, California, United States